CLINICAL TRIAL: NCT01025999
Title: Mechanisms of Glycemic Improvement After Gastrointestinal Surgery
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David Flum, Professor, University of Washington
Other Study IDs: 36417-A; 1R01DK084324-01 (NIH)
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus, Type II
Keywords: RYGB; Gastrostomy tube; DM; Gastric Bypass
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma collected to measure markers of metabolic activity.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- RYGB: UWMC patients undergoing RYGB surgery with routine placement of Gastrostomy tube.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
This study is designed as a prospective clinical trial aimed at investigating the mechanisms behind observed improvements in type 2 diabetes mellitus (T2DM) following bariatric surgery. The majority of patients with T2DM who are undergoing Roux-en-Y gastric bypass (RYGB) surgery, in particular, experience complete remission of T2DM almost immediately post-surgery. This response occurs before significant weight loss is possible. To assess the mechanisms involved with disease resolution, the investigators propose a study to evaluate patients at the UW Medical Center (UWMC) who have T2DM and are undergoing RYGB with G (gastronomy)-tube placement as part of their clinical care. The investigators are interested in this sub-population as the G-tube allows us the unique opportunity to evaluate glycemic control and insulin response following delivery or exclusion of nutrients to the otherwise bypassed portion of the gastrointestinal tract. The investigators hypothesize that nutrient delivery to the proximal GI tract will reverse RYGB-mediated improvements in glucose homeostasis, possibly in association with changes in nutrient-regulated gut peptides involved in glucose control.

DETAILED DESCRIPTION:
Roux-en-Y gastric bypass surgery causes complete, durable remission of type 2 diabetes (T2DM) in 84% of cases, typically within a few days to weeks after surgery. Mounting evidence indicates that this dramatic phenomenon results from effects beyond those related to weight loss and reduced caloric intake alone. The mechanisms mediating the weight-independent anti-diabetes impact of RYGB are unknown, and elucidating them could lead to new diabetes medicines. Human subjects will undergo frequently sampled I.V. glucose tolerance tests (FS-IVGTT) and tracer-enhanced hyperinsulinemic/euglycemic clamps (to measure insulin secretion and sensitivity) before RYBG and 3 times in the first six weeks afterward, during which the proximal small bowel will either be excluded from nutrient contact or exposed to nutrients delivered through an indwelling gastric cannula. We hypothesize that nutrient delivery to the proximal GI tract will reverse RYGB-mediated improvements in glucose homeostasis, possibly in association with changes in nutrient-regulated gut peptides involved in glucose control. Our study will allow us to test the upper intestinal hypothesis rigorously in man, and whether the hypothesis is confirmed or refuted, we will gain valuable new insights into the mechanisms of improved glucose control early after RYGB.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater and planning to undergo RYGB at UWMC
* Ability to speak English and communicate effectively with research staff
* Ability to return for follow-up visits at UWMC
* Adequate IV access
* A G-tube is planned as part of the bariatric surgical procedure
* Documented T2DM (fasting plasma glucose >125 mg/dL) that is treated with lifestyle efforts or by taking acceptable oral medications

Exclusion Criteria:

* Informed consent not obtained
* Unlikely to comply with the protocol
* Current HbA1c >8.5% or fasting blood glucose >180 mg/dL
* Serum creatinine >1.7 mg/dL
* Use of unacceptable diabetes medications at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planning to undergo RYGB at UWMC with planned placement of gastrostomy tube.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Determine if the improvements in glycemic control occurring early after RYGB can be reversibly inactivated and activated through delivery or exclusion of nutrients in the bypassed proximal small intestine. | 1/2010 - 6/2014

SECONDARY OUTCOMES:
To evaluate whether improvements in glucose control occurring early after RYGB are related to altered insulin secretion, insulin sensitivity, or both. | 1/2010-6/2014

CONTACTS AND LOCATIONS:
Overall Officials: David R Flum, MD, MPH, Principal Investigator — University of Washington; David E Cummings, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States